CLINICAL TRIAL: NCT01919970
Title: Exposure-Focused Family-Based CBT for Youth With ASD and Comorbid Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-FET 2013
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Autism; Asperger's Syndrome; Pervasive Developmental Disorder Not Otherwise Specified; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder; Obsessive-compulsive Disorder; Specific Phobia
Keywords: Autism; Asperger's Syndrome; Pervasive Developmental Disorder Not Otherwise Specified; Treatment; Cognitive-behavioral therapy; Anxiety; Children; Therapy; Generalized Anxiety Disorder; Social Phobia; Separation Anxiety Disorder; Obsessive-compulsive Disorder; Specific Phobia
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Obsessive-Compulsive Disorder; Phobia, Specific; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy Condition (Experimental): This arm is the experimental condition; it consists of 12 weekly CBT sessions. The therapy protocol will begin with an introductory education session which will include development of a fear hierarchy, followed by 11 sessions of in vivo exposures to feared triggers.
  Interventions: Other: Cognitive Behavioral Therapy
- Treatment as Usual (Active Comparator): This arm acts as the comparison condition. Participants randomized to this arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice; and will be monitored through periodic study assessment.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — This condition involves 12 weekly CBT sessions.
  Arms: Cognitive Behavioral Therapy Condition
Other: Treatment as usual — This condition allows participants to seek out various services. Considering the number of possible treatment options, there is no way to identify or list them.
  Arms: Treatment as Usual

SUMMARY:
Autism spectrum disorders affect as many as 1 out of 88 children and are related to significant impairment in social, adaptive, and school functioning. Co-occurring conditions, such as anxiety, are common and may cause substantial distress and impairment beyond that caused by the autism diagnosis. Accordingly, we are proposing a randomized controlled trial to examine the effectiveness of a form of cognitive-behavioral therapy relative to treatment as usual (TAU) in 50 youth ages 6-12 with autism spectrum disorders and comorbid anxiety.

DETAILED DESCRIPTION:
Autism spectrum disorders affect as many as 1 out of 88 children and are related to significant impairment in social, adaptive, and school functioning. Co-occurring conditions, such as anxiety, are common and may cause substantial distress and impairment beyond that caused by the autism diagnosis. Many children with anxiety disorders, especially those on the autism spectrum, do not receive evidence based treatment, which has fueled the development and evaluation of cognitive-behavioral therapy (CBT). Accordingly, we are proposing a randomized controlled trial to examine the efficacy of exposure based CBT that heavily incorporates parents (EF-CBT) relative to a TAU condition (TAU) in 50 youth ages 6-12 years with ASD and comorbid anxiety disorder(s).

ELIGIBILITY:
Inclusion Criteria:

* Outpatient children with an autism spectrum disorder between the ages 6-12 years.
* Meets criteria for a diagnosis of one of the following anxiety disorders: generalized anxiety disorder, separation anxiety disorder, social phobia, specific phobia, panic disorder or obsessive-compulsive disorder.
* Minimum score of 12 on the Pediatric Anxiety Rating Scale - Severity Scale.
* Child has a Full Scale and Verbal Comprehension IQ > 80.

Exclusion Criteria:

* Current clinically significant suicidality or engagement in suicidal behaviors within the last 6 months.
* Presence of any clinical features requiring a higher level of care (inpatient or partial hospital treatment).
* Any lifetime diagnosis (meeting DSM-IV criteria) of bipolar disorder, schizophrenia or schizoaffective disorder; or Substance abuse in the past 6 months.
* Initiation of an antidepressant medication within 10 weeks before study enrollment or an antipsychotic medication 6 weeks before study enrollment or the child has changed the dose of an established medication within 6 weeks before study enrollment (4 weeks for antipsychotic) or during psychotherapy (unless the dose is lowered because of side effects). If the child is on a medication, she or he can remain on it at its current dose. While in their treatment arm, children randomized to the EF-CBT condition will not be able to continue or initiate psychosocial interventions targeting anxiety(psychotherapy, certain types of social skills training, applied behavior analysis targeting anxiety). Those in the TAU arm will be able to seek out psychiatric/psychological services at their discretion.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Center for Neuropsychiatry, St. Petersburg, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 32 subjects were enrolled in this study (versus the N=40) indicated in the Protocol attached.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Started | 14 | 18
Completed | 11 | 18
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 18 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.07 (2.89) | 10 (2.83) | 10.03 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 10 | 16 | 26
Region of Enrollment [Number; unit: participants]
  United States | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale
Description: This scale measures the severity of anxiety symptoms in children. The total scale range is 0-30 where 0 is the minimum and 30 the maximum. Higher scores correspond to more severe anxiety symptom severity. The total scale was used which corresponds to summing the 6 severity items.
  The outcome measure is reporting a change score in which the score at baseline is compared to the score at 12 weeks (post-treatment). This is analyzed as a function of groups/condition (cognitive behavioral therapy versus Treatment as Usual).
Time Frame: After an average of 12 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Number analyzed (Participants) | 14 | 18
units on a scale | 7.79 (5.37) | 15.06 (3.21)

2. Secondary Outcome: Clinical Global Impression - Severity Scale
Description: This scale measures the severity of anxiety symptoms in children. The total scale range is 0-6 where 0 is the minimum and 6 the maximum. Higher scores correspond to more severe anxiety symptom severity. The scale consists of only 1 item that a clinician rates based on their judgement of anxiety severity.
  The outcome measure is reporting a change score in which the score at baseline is compared to the score at 12 weeks (post-treatment). This is analyzed as a function of groups/condition (cognitive behavioral therapy versus Treatment as Usual).
Time Frame: After an average of 12 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
Number analyzed (Participants) | 14 | 18
units on a scale | 2.25 (.87) | 3.67 (.69)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Cognitive Behavioral Therapy Condition | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18

LIMITATIONS AND CAVEATS:
Small sample size. Short follow-up period. Many youth receiving usual care did not seek active treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No